CLINICAL TRIAL: NCT06901908
Title: Role of Cytomorphometry and BRAFV600E Immunocytochemistry With a Cytologic Diagnosis "Suspicious for Papillary Thyroid Carcinoma"
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salwa Mohamed, Principal Investigator, Assiut University
Other Study IDs: FNACSTUDY
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Suspicious for Papillary Thyroid Carcinoma
Keywords: fine needle aspiration; suspicious for malignancy; suspicious for papillary thyroid carcinoma; BRAFV600E; cytomorphometry; thyroid gland
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — FNAC smears diagnosed as suspicious for papillary thyroid carcinoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Thyroid nodules (TNs) are a common finding, detected by ultrasound in about 70% of healthy individuals, with women being four times more affected. While most TNs are benign, the primary clinical goal is to exclude malignancy, which occurs in 4-6.5% of cases. Risk factors for TNs include age, gender, iodine imbalance, family history, and radiation exposure. Thyroid cancer incidence has risen due to improved diagnostic methods such as ultrasound, FNAC, CT, MRI, and PET scans.

Papillary thyroid carcinoma (PTC) is the most common thyroid malignancy (90%), followed by follicular, Hurthle cell, medullary, and anaplastic carcinomas. Most thyroid cancers have an excellent prognosis, with a 5-year survival rate of 98.6%. FNAC is the gold standard for diagnosing TNs, and the Bethesda system (TBSRTC) categorizes cytology results into six groups with varying malignancy risks. The "suspicious for malignancy" category (74% risk) includes mostly suspicious papillary thyroid carcinoma (SPTC), but false positives occur, especially in cases of Hashimoto's thyroiditis.

SPTC diagnosis can be challenging, leading to potential overtreatment. To improve diagnostic accuracy, additional techniques like detailed ultrasonographic criteria, intraoperative frozen section, and molecular marker testing are used. Cytomorphometric analysis has been explored for distinguishing benign from malignant thyroid lesions, assessing nuclear size, shape, and chromatin patterns. Most studies have focused on histological sections, but applying morphometry to cytology could enhance automated and accurate diagnoses.

Molecular studies reveal that PTCs primarily arise from MAPK pathway mutations, with BRAFV600E being the most common (60%). This mutation is strongly associated with aggressive tumor behavior and recurrence. BRAFV600E testing combined with FNAC significantly improves diagnostic accuracy, increasing sensitivity from 76.71% (mutation testing alone) to 96.62% when combined with cytology. This integration has reduced false-negative PTC diagnoses and facilitated targeted therapies.

DETAILED DESCRIPTION:
Thyroid nodules are common clinical finding in routine daily medical and surgical practice. They are discovered by ultrasonography in about 70% of clinically healthy individuals. Thyroid nodules are four times more prevalent in women and up to 90% of cases are caused by benign conditions.

The main target of clinical management of thyroid nodules is exclusion of malignancy (4-6.5% of all thyroid nodules), assessment of pressure symptoms and evaluation of thyroid dysfunction .

Many risk factors were identified related to development of thyroid nodules including advanced age, gender, increased or decreased iodine, family history of cancer or polyposis and history of head and neck radiation. The most common thyroid nodules are colloid nodules, Hashimoto's thyroiditis, subacute thyroiditis, cysts, follicular adenoma and thyroid cancers.

Regarding thyroid malignant tumors, the incidence of thyroid cancer increased over the past decades in the United States and internationally. It's the 7th most common cancer in the general population and the 5th most common in women. The incidence of thyroid cancer is about 3 times higher in women than men and it increases from adolescence to middle age with the peak around 55 years in women and 65 years in men then decreasing with older age.

The increase of number of cancer cases is caused by increased diagnosis resulting from the widespread use of diagnostic tools including ultrasonography imaging, fine needle aspiration cytology , computed tomography , magnetic resonance imaging and fluorodeoxyglucose positron emission tomography. In addition to the increase in the exposure to the etiologic factors as ionizing radiation during childhood and obesity.

Papillary thyroid carcinoma (PTC) is the most common histologic type of thyroid cancers representing 90% of cases. The remaining 10% include follicular thyroid carcinoma 4%, Hurthle cell carcinoma 2%, medullary thyroid carcinoma 2% and anaplastic thyroid carcinoma 1% .

The prognosis of thyroid cancer is excellent because most cases are papillary thyroid carcinomas localized to the thyroid gland during diagnosis. The 5-year survival rate is 98.6% overall, 99.9% for localized, 98.3% for regional and 54.9% for distant metastasis .

Fine-needle aspiration cytology (FNAC) of the thyroid gland is a gold standard accurate diagnostic test routinely used in the initial evaluation of thyroid nodules as it is simple, safe, cost-effective and has favorable accuracy. The sensitivity and specificity of thyroid FNAC are 68-98% and 56-100% respectively with failure rates are because of the technique and experience of the performance .

The Bethesda system for reporting thyroid cytopathology (TBSRTC) was first published in 2010 and updated many times to standardize reporting terminology and for better communication between cytopathologists and clinicians.

The 2023 Bethesda system for reporting thyroid cytopathology is a simple category-based reporting system for fine needle aspiration cytology (FNAC) of thyroid and became one of the most used reporting and diagnostic methods and includes 6 categories.

Category (I) non diagnostic with 13%(5-20) risk of malignancy, Category (II) benign with 4%(2-7) risk of malignancy, Category (III) atypia of undetermined significance with 22%(13-30) risk of malignancy, Category (IV) follicular neoplasm with 30%(23-34) risk of malignancy, Category (V) suspicious for malignancy with 74%(67-83) risk of malignancy and Category (VI) malignant with 97%(97-100) risk of malignancy.

The suspicious for malignancy category is used when cytomorphologic features is inconclusive and raise a strong suspicion of malignancy but are quantitatively or qualitatively insufficient for a conclusive diagnosis and the usual management in this case is molecular testing, lobectomy or near total thyroidectomy.

The suspicious for malignancy (SFM) according to Bethesda system category includes suspicious for papillary thyroid carcinoma (SPTC) which is the most common subtype (more than 90%) and less frequently suspicious for non-papillary carcinoma which consists of suspicious for medullary thyroid carcinoma, suspicious for malignant lymphoma, suspicious for poorly differentiated carcinoma and suspicious for malignancy not otherwise specified.

Suspicious for papillary thyroid carcinoma is diagnosed due to patchy nuclear changes (unremarkable follicular cells admixed with cells showing nuclear enlargement, pallor, grooves and fine chromatin, scant or absent intranuclear pseudoinclusions and absent papillary architecture) , incomplete nuclear changes (generalized nuclear enlargement, pallor and grooves, scant or absent irregular nuclear membrane and intranuclear pseudoinclusions and absent papillary architecture and psammoma bodies), sparsely cellular specimen or cystic degeneration (background of cystic debris and macrophages, nuclear enlargement and pallor, atypical histocytoid cells with cytoplasmic vacuoles and absent papillary architecture and psammoma bodies.

Suspicious for papillary thyroid carcinoma is diagnosed in 2.4-8% of fine needle aspiration results and 60-80% of them are confirmed in resected specimens to be papillary thyroid carcinoma and the rest of cases showed benign conditions as chronic lymphocytic thyroiditis (Hashimoto thyroiditis) and nodular hyperplasia. Hashimoto thyroiditis is one of the most common factors in false positive papillary thyroid carcinoma diagnosis because of the strong overlap of morphological features between them.

Suspicious for papillary thyroid carcinoma diagnosis is confusing for surgeons and patients and makes the optimal surgical decision difficult as the prevalence of malignancy in this diagnostic category is high. Some surgeons proceed for total thyroidectomy and this makes about 25% of patients (false positive cases) may suffer from oversurgery and in need for hormone replacement therapy for life. Many trials were made to increase the accuracy of detection of malignancy in this category and decrease the possibility of oversurgery. Some authors applied detailed ultrasonographic criteria for cases diagnosed cytologically as suspicious for papillary thyroid carcinoma and reported increase of accuracy from 86% to 94% while others performed intraoperative frozen section and ancillary tests as molecular markers.

Cytomorphometric analysis has been used as a clinical diagnostic tool and discussed in the literature for over 30 years. It has been used in many organs like nasopharynx, skin, urinary bladder, colon, breast and thyroid. Morphometry is computerized procedure performed through the quantitative analysis of geometric features of structures with any dimension. The nuclear morphometry of malignant nuclei including the size, shape, and chromatin pattern, are different from those of nonmalignant cell nuclei, which allows nuclear morphometry to distinguish between benign and malignant cases. Using nuclear morphometry, we can quantify a number of parameters such as those related to nuclear size and shape.

Morphometry can help as an adjunct to morphological features in thyroid lesions when correctly applied with appropriate cutoffs. Till now, majority of image analysis studies have been performed on histopathological sections and only few studies performed on cytological smears. It has been suggested that nuclear morphometric parameters such as nuclear area and perimeter and shape factors may allow differentiation between thyroid lesions. Applying morphometry to cytology would be useful for the purpose of automated morphometric screening as well as accurate diagnosis of thyroid tumors.

The computerized morphometric study of thyroid histological slides identified efficient morphometric parameters that distinguish the differences between benign and malignant epithelial cells and the most reliable parameters are area, perimeter, length, width, the degree of roundness and irregularity of the nuclear membranes.

A study revealed that the cytomorphometric image analysis with cytomorphology has the potential for distinguishing not only the benign, follicular neoplasm/suspicious for a follicular neoplasm, malignant thyroid lesions of Bethesda system but also can distinguish nodules with follicular patterns as follicular variant of papillary carcinoma, follicular adenoma and follicular carcinoma.

Many molecular based analytic studies have proved that most papillary thyroid carcinomas are caused by two distinct signaling mechanisms of the MAPK ( Mitogen-activated protein kinase) pathway, either BRAF-like or RAS-like.

The most common gene mutation in papillary thyroid carcinoma (60%) is a missense mutation in the BRAF oncogene, valine (V) substituting glutamic acid (E) at amino acid position 600, which finally drives mitogen-activated protein kinase pathway signaling.

A systematic review and meta-analysis showed that the recurrence rate in BRAFV600E mutated papillary thyroid carcinomas (24.9%) was two times high as wild-type papillary thyroid carcinomas (12.6%). The BRAFV600E mutated PTCs has more risk for lymph node metastasis, extrathyroidal extension and associated with advanced AJCC III/IV stage.

The access to molecular testing has facilitated the use of therapeutic agents targeting specific mutations as BRAFV600E.

The BRAFV600E mutation is very common in papillary thyroid carcinoma (38-90% incidence) and rarely present in benign thyroid lesions so its diagnostic specificity is high. It leads to abnormal activation of the mitogen-activated protein kinase pathway which plays an important role in the development of papillary thyroid carcinoma . It was reported that fine needle aspiration cytology combined with the preoperative BRAFV600E mutation detection can improve the diagnostic performance for thyroid nodules compared to fine needle aspiration cytology alone.

The sensitivity and specificity of the BRAFV600E mutation testing alone for papillary thyroid carcinoma were 76.71% and 100% respectively and increased to 96.62% and 88.03% respectively when combined with cytology. So, the combination between fine needle aspiration cytology and BRAFV600E mutation tests has decreased the false negatives in papillary thyroid carcinoma diagnosis.

Material and methods:

A retrospective descriptive study will be performed on FNA smears of thyroid nodules received in the Department of Pathology at Assiut University Hospital over a six-year period (2018-2025). The study will review Papanicolaou (PAP) and Hematoxylin & Eosin (H&E) stained smears from 45 patients with thyroid nodules diagnosed as suspicious for papillary thyroid carcinoma (Bethesda V), combined with the histopathological data of their resected thyroid specimens.

All clinical, radiological and pathological data will be collected from medical records.

Personal data including age and gender, clinical data as number of thyroid nodules and their size and the presence or absence of cervical lymph node enlargement and pressure symptoms and radiological data as thyroid imaging reporting and data system (TI-RADS) which includes composition, echogenicity, shape, margin and punctate echogenic foci will be collected.

Morphometric study:

For each case, 50 nuclei from follicular cells within the suspicious cellular group, with well-preserved morphology, will be selected. Nuclei that will exhibit overlapping, will be obscured by inflammation, blood, or mucin, or will display degenerative changes will be excluded. Preference will be given to isolated nuclei or those just touching each other without overlap with a clean background. Each selected nucleus focused on using a 1000x oil immersion objective lens will be imaged using a digital camera and will be analyzed with Image Analysis Software. The software will assign a specific number to each nucleus in the image and quantify its morphometric parameters.

Immunocytochemical study:

BRAFV600E immunocytochemistry will be applied on the smears after destaining them.

Smears will be stained with BRAFV600E antibodies with immunoperoxidase staining as a visualization method.

Antibody dilution and incubation time will be conducted according to manufacturer's instructions.

Correlation between results of cytomorphometric studies, results of BRAFV600E mutation tests and the results of histopathological slides will be done.

ELIGIBILITY:
Inclusion Criteria:

* Only Papanicolaou (PAP) and Hematoxylin & Eosin (H&E) stained FNAC smears diagnosed as suspicious for papillary thyroid carcinoma will be included in the study.
* Only FNAC smears with well-preserved nuclear morphology will be included in the study.
* Smears with histopathological slides.

Exclusion Criteria:

* FNAC smears lacking histopathological confirmation.
* Smears with extensive nuclear overlap and poor morphology.
* Smears obscured by inflammation, blood, or mucoid material.
* Smears exhibiting cellular degenerative changes or drying artifacts.
* Any patient with missing data.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Only Papanicolaou (PAP) and Hematoxylin & Eosin (H&E) stained FNAC smears with well-preserved nuclear morphology and diagnosed as suspicious for papillary thyroid carcinoma will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Role of Cytomorphometry and BRAFV600E Immunocytochemistry with a Cytologic Diagnosis "Suspicious for Papillary Thyroid Carcinoma" | 3 months
  * To evaluate the risk of malignancy in TNs diagnosed as SPTC by FNAC.
  * To characterize the different morphometric parameters in cases diagnosed cytologically as SPTC.
  * To evaluate the immunocytochemical expression of BRAFV600E in cases diagnosed cytologically as SPTC.
  * To evaluate the utility of cytomorphometric analysis and BRAFV600E immune-staining alone or in combination in upgrading the diagnostic accuracy of SPTC cases.

CONTACTS AND LOCATIONS:
Overall Officials: Nermeen A Kamel, Principal Investigator — Assiut Univesity

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhu Y, Ren W, Song Y, Fan Z, Wang Q, Jin H, Guo Y, Bai Y. Cytomorphologic features as predictors of aggressiveness in patients with pT1 papillary thyroid carcinoma: a retrospective study of associations with clinicopathological parameters in 226 fine-needle aspirates. Gland Surg. 2021 Jan;10(1):319-327. doi: 10.21037/gs-20-618. PMID 33633988
- [Background] Tamhane S, Gharib H. Thyroid nodule update on diagnosis and management. Clin Diabetes Endocrinol. 2016 Oct 3;2:17. doi: 10.1186/s40842-016-0035-7. eCollection 2016. PMID 28702251
- [Background] Priya SS, Sundaram S. Morphology to morphometry in cytological evaluation of thyroid lesions. J Cytol. 2011 Jul;28(3):98-102. doi: 10.4103/0970-9371.83462. PMID 21897541
- [Background] Parker KG, White MG, Cipriani NA. Comparison of Molecular Methods and BRAF Immunohistochemistry (VE1 Clone) for the Detection of BRAF V600E Mutation in Papillary Thyroid Carcinoma: A Meta-Analysis. Head Neck Pathol. 2020 Dec;14(4):1067-1079. doi: 10.1007/s12105-020-01166-8. Epub 2020 May 1. PMID 32358715
- [Background] Mohorea I, Socea B, Carap AC, Serban D, Ceausu Z, Ceausu M. Morphometric study in thyroid tumors. Exp Ther Med. 2023 Sep 6;26(4):497. doi: 10.3892/etm.2023.12196. eCollection 2023 Oct. PMID 37745041
- [Background] Mahajan A, Lin X, Nayar R. Thyroid Bethesda reporting category, 'suspicious for papillary thyroid carcinoma', pitfalls and clues to optimize the use of this category. Cytopathology. 2013 Apr;24(2):85-91. doi: 10.1111/j.1365-2303.2012.00966.x. Epub 2012 Feb 22. PMID 22356185
- [Background] Leiker AJ, Yen TW, Cheung K, Evans DB, Wang TS. Cost analysis of thyroid lobectomy and intraoperative frozen section versus total thyroidectomy in patients with a cytologic diagnosis of "suspicious for papillary thyroid cancer". Surgery. 2013 Dec;154(6):1307-13; discussion 1313-4. doi: 10.1016/j.surg.2013.06.031. PMID 24238049
- [Background] Kwak JY, Kim EK, Kim MJ, Hong SW, Choi SH, Son EJ, Oh KK, Park CS, Chung WY, Kim KW. The role of ultrasound in thyroid nodules with a cytology reading of "suspicious for papillary thyroid carcinoma". Thyroid. 2008 May;18(5):517-22. doi: 10.1089/thy.2007.0271. PMID 18407756
- [Background] Kitahara CM, Schneider AB. Epidemiology of Thyroid Cancer. Cancer Epidemiol Biomarkers Prev. 2022 Jul 1;31(7):1284-1297. doi: 10.1158/1055-9965.EPI-21-1440. No abstract available. PMID 35775227
- [Background] Khatri P, Choudhury M, Jain M, Thomas S. Role of morphometry in the cytological differentiation of benign and malignant thyroid lesions. J Cytol. 2017 Jan-Mar;34(1):1-4. doi: 10.4103/0970-9371.197579. PMID 28182069
- [Background] Kezlarian B, Lin O. Artificial Intelligence in Thyroid Fine Needle Aspiration Biopsies. Acta Cytol. 2021;65(4):324-329. doi: 10.1159/000512097. Epub 2020 Dec 16. PMID 33326953
- [Background] Kant R, Davis A, Verma V. Thyroid Nodules: Advances in Evaluation and Management. Am Fam Physician. 2020 Sep 1;102(5):298-304. PMID 32866364
- [Background] Jing X, Michael CW. Potential pitfalls for false suspicion of papillary thyroid carcinoma: a cytohistologic review of 22 cases. Diagn Cytopathol. 2012 May;40 Suppl 1:E74-9. doi: 10.1002/dc.21726. Epub 2011 May 11. PMID 21563322
- [Background] Fu J, Yin X, Wang X, Xiao S, Wu X, Duan C, Yu W, Zhang G. Diagnostic value of FNAC combined with BRAFV600E mutation detection in Hashimoto's thyroiditis complicated with papillary thyroid carcinoma. Front Endocrinol (Lausanne). 2024 May 16;15:1366724. doi: 10.3389/fendo.2024.1366724. eCollection 2024. PMID 38818506
- [Background] Chowsilpa S, Jones R, Hang JF, Ali SZ. Characterization of "suspicious for malignancy" for non-papillary carcinoma diagnoses on thyroid fine-needle aspiration. J Am Soc Cytopathol. 2021 Mar-Apr;10(2):148-154. doi: 10.1016/j.jasc.2020.06.007. Epub 2020 Jul 15. PMID 32773337
- [Background] Chen H, Song A, Wang Y, He Y, Tong J, Di J, Li C, Zhou Z, Cai X, Zhong D, Da J. BRAFV600E mutation test on fine-needle aspiration specimens of thyroid nodules: Clinical correlations for 4600 patients. Cancer Med. 2022 Jan;11(1):40-49. doi: 10.1002/cam4.4419. Epub 2021 Dec 1. PMID 34851044
- [Background] Chaurasia JK, Ilyas AM, Walke V, Gupta V, Kapoor N. The Role of Cytomorphometric Image Analysis in the Diagnosis of Thyroid Nodules. Cureus. 2023 Apr 20;15(4):e37872. doi: 10.7759/cureus.37872. eCollection 2023 Apr. PMID 37214005
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- [Background] AlSaedi AH, Almalki DS, ElKady RM. Approach to Thyroid Nodules: Diagnosis and Treatment. Cureus. 2024 Jan 13;16(1):e52232. doi: 10.7759/cureus.52232. eCollection 2024 Jan. PMID 38352091
- [Background] Ali SZ, Baloch ZW, Cochand-Priollet B, Schmitt FC, Vielh P, VanderLaan PA. The 2023 Bethesda System for Reporting Thyroid Cytopathology. Thyroid. 2023 Sep;33(9):1039-1044. doi: 10.1089/thy.2023.0141. Epub 2023 Jul 8. PMID 37427847